CLINICAL TRIAL: NCT05281263
Title: A Phase 1 Trial of the Safety, Tolerability, and Immunogenicity of BLB-201 Vaccine in Healthy Young Adults and Older Adults
Brief Title: Phase 1 Study of BLB-201 Vaccine in Healthy Young and Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blue Lake Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BLB-201-001
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Human respiratory syncytial virus (RSV); lower respiratory tract infection (LRTI)
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1, young adult cohort (age 18-59) (Experimental): BLB-201 administered as a single dose of 10^7.5 PFU by intranasal route on Day 1
  Interventions: Biological: CPI-RSV-F Vaccine (BLB-201)
- Group 2, older adult cohort (age 60-75) (Experimental): BLB-201 administered as a single dose of 10^7.5 PFU by intranasal route on Day 1
  Interventions: Biological: CPI-RSV-F Vaccine (BLB-201)

INTERVENTIONS:
Biological: CPI-RSV-F Vaccine (BLB-201) — see arm/group description

SUMMARY:
This Phase 1 trial is an open-label trial to evaluate the safety, tolerability and immunogenicity of a single dose (10^7.5 PFU) of intranasal BLB-201 (a recombinant parainfluenza virus type 5) administered as a single dose in 15 healthy young adults ages 18-59 years, and 15 older adults ages 60-75 years.

DETAILED DESCRIPTION:
This will be an open-label, age-escalation phase 1 trial of the PIV5 virus-vectored BLB-201 vaccine in healthy adults (males and nonpregnant females) 18 to 59 years of age (Group 1), and 60 to 75 years of age (Group 2). The trial is designed to assess the safety, tolerability, and immunogenicity of a single dose of intranasal BLB-201 at 10^7.5 plaque- forming units (PFU) in both Group 1 and Group 2. The first 4 subjects in each group will be enrolled as sentinels and vaccination will proceed in a staged fashion.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent prior to initiation of any trial procedures.
* Be able to understand and agrees to comply with planned trial procedures and be available for all trial visits and phone calls.
* Healthy male or non-pregnant female, between 18 and 59 years of age (Group 1) or between60 and 75 years of age (Group 2), inclusive, at time of trial vaccination.
* Women of childbearing potential must agree to use or have practiced true abstinence or use at least one acceptable primary form of contraception. Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).
* Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to each vaccination.
* Male subjects of childbearing potential* must use condoms to ensure effective contraception with a female partner of childbearing potential from vaccination until 90 days after vaccination. Such female partners must also use an acceptable form of primary contraception as described under inclusion criterion #4. If barrier methods are to be used, then double barrier methods of protection are required, i.e. male condom, in combination with a cap, diaphragm, or sponge with spermicide. *Biological males who are post-pubertal and considered fertile until permanently sterile by bilateral orchiectomy or vasectomy.
* Male subjects agree to refrain from sperm donation from the time of vaccination until 90 days after vaccination.
* Female subjects agree to refrain from egg donation from time of vaccination until 90 days after vaccination.
* In good health.

Exclusion Criteria:

* History of clinically-significant or major disease that may interfere with a subject completing the trial and necessary investigations.
* Have an acute illness as determined by the site PI or sub-investigator within 72 hours prior to trial vaccination.
* Women who are pregnant, lactating, or unwilling to take effective measures to prevent pregnancy for at least 3 months after vaccination.
* Receipt of any live vaccine within the 30 days prior to trial vaccination.
* Receipt of any inactivated vaccine within the 14 days prior to trial vaccination.
* Receipt of any investigational vaccine within 12 months prior to trial vaccination (not including vaccines made available under an FDA emergency-use authorization).
* Any prior receipt of any investigational RSV vaccine or any PIV5-based vaccine (e.g. CVXGA1).
* Intention to receive any other vaccination before the last in person scheduled visit of the trial.
* Receipt or anticipated receipt of immunoglobulin or blood products within 90 days prior to trial vaccination through trial period.
* Loss (including blood donations) of 470 mL or more of blood within 90 days prior to trial vaccination.
* Receipt or anticipated receipt of systemic glucocorticoids within 30 days prior to trial vaccination through trial period.
* Receipt or anticipated receipt of any antiviral drug within 7 days prior to vaccination through 14 days after trial vaccination.
* History and/or symptoms indicative of upper or lower respiratory tract infection within 14 days prior to initial trial vaccination (e.g. cough, sore throat, body temperature of 99.5°F or greater, nasal congestion, dyspnea, tachypnea, wheezing, fatigue, myalgia).
* Any clinically significant history of heavy nosebleeds.
* History of chronic sinus infection.
* Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
* History of postinfectious or postvaccine neurological sequelae.
* Autoimmune, inflammatory, vasculitic, or rheumatic disease or immunodeficiency disorder.
* Any significant abnormality altering the anatomy of the nose.
* History of significant/severe wheeze, respiratory symptoms resulting in hospitalization, or known bronchial hyperreactivity to viruses.
* History of asthma or reactive airway disease as an adult, cystic fibrosis, bronchopulmonary dysplasia, or chronic obstructive pulmonary disease.
* History of anaphylaxis or other severe allergic reaction, e.g., generalized urticaria, angioedema, or other significant reaction to any previous licensed or unlicensed vaccines. - Have a diagnosis of schizophrenia, bipolar disease, or other psychiatric disease that may interfere with subject compliance or safety evaluations.
* Use or anticipated use during the conduct of the trial of high-dose inhaled corticosteroids from 30 days prior to 14 days after trial vaccination.
* Receipt or anticipated receipt of, within 7 days prior to through 28 days after trial vaccination, any intranasal medication including FDA-approved prescription or over-the-counter products or non-FDA-approved alternative medicine products (e.g. Ayurvedic oil or other naturopathic substances).
* Currently smoking or vaping, or history of regular smoking or vaping in the past two years.
* Anticipated use of nasal irrigation (e.g. Neti Pot™) after enrollment through 28 days after trial vaccination.
* Positive hepatitis C or HIV serology, or positive hepatitis B serology not attributable to hepatitis B immunization.
* History of alcohol or drug abuse within 5 years prior to trial vaccination.
* Received experimental agent within 30 days prior to trial vaccination or expects to receive experimental agent (not including vaccines made available under an FDA emergency use authorization) anytime during the 6-month trial period.
* Female subjects that are breastfeeding or plan to breastfeed during the trial.
* Subjects who reside in a nursing home.
* Any condition that would in the opinion of the site investigator place the subject at unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Solicited Adverse Events | Day 1-8
  Frequencies and grades of solicited local and systemic AEs during a 7-day period after dosing.
Unsolicited Adverse Events | Day 1-29
  Frequencies and grades of unsolicited AEs during a 28-day period after dosing.

SECONDARY OUTCOMES:
Serum IgG titers to RSV protein | Day 15, and Day 29
  Change in RSV specific IgG titers after the first dose of BLB-201.
Serious Adverse Events through trial completion | Day 1-181
  Frequencies of Serious Adverse Events (SAEs) categorized by vaccine relatedness from the first dose of BLB-201 through trial completion (approximately 6 months after dosing).
Serious adverse events, new-onset chronic medical conditions, and adverse events of special interest | Day 1-181
  Frequencies of Serious Adverse Events (SAEs) categorized by vaccine relatedness, new-onset chronic medical conditions (NOCMCs), and adverse events of special interest (MAAEs), from the first dose of BLB-201 through trial completion (approximately 6 months after dosing).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Spearman, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD underlying the results reported in any published articles (text, tables, figures, appendices) will be shared.
Supporting Information: Study Protocol
Time Frame: 5 years, beginning as soon as possible (but no later than 12 months) after article publication.
Access Criteria: Data will be made available to investigators and institutions upon request. Requests should be directed to the CyanVac authors of the publication(s).

REFERENCES:
- [Result] Spearman P, Jin H, Knopp K, Xiao P, Gingerich MC, Kidd J, Singh K, Tellier M, Radziewicz H, Wu S, McGregor M, Freda B, Wang Z, John SP, Villinger FJ, He B. Intranasal parainfluenza virus type 5 (PIV5)-vectored RSV vaccine is safe and immunogenic in healthy adults in a phase 1 clinical study. Sci Adv. 2023 Oct 27;9(43):eadj7611. doi: 10.1126/sciadv.adj7611. Epub 2023 Oct 25. PMID 37878713